CLINICAL TRIAL: NCT02450526
Title: A Phase III, Randomised, Double Blind and Open Label Phase, Multicentre, Active and Placebo Controlled Study to Investigate the Efficacy and Safety of Dysport Including a Comparison to Botox in the Treatment of Moderate to Severe Glabellar Lines, and to Assess the Long Term Efficacy and Safety of Dysport Following Repeated Treatments in This Indication
Brief Title: Dysport in the Treatment of Glabellar Lines in Chinese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Y-52-52120-158
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AbobotulinumtoxinA (Experimental): Dysport, 50 Units, divided into five injections into the glabellar area. Administered in double blind fashion at cycle 1 followed by up to 4 cycles Dysport, 50 Units administered with an interval period depending on response, no less than 12 weeks between each treatment cycle.
  Interventions: Biological: Botulinum toxin type A
- OnabotulinumtoxinA (Active Comparator): Botox will be administered in treatment cycle 1 only. On Day 1, 20 Units, divided into five injections into the glabellar area.
  Interventions: Biological: Botulinum toxin type A
- AbobotulinumtoxinA Placebo (Placebo Comparator): Dysport placebo will be administered in treatment cycle 1 only. On Day 1, 50 Units, divided into five injections into the glabellar area.
  Interventions: Drug: Placebo
- OnabotulinumtoxinA Placebo (Placebo Comparator): Botox placebo will be administered in treatment cycle 1 only. On Day 1, 20 Units, divided into five injections into the glabellar area.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: AbobotulinumtoxinA
Biological: Botulinum toxin type A
  Other Names: OnabotulinumtoxinA (Botox®)
  Arms: OnabotulinumtoxinA
Drug: Placebo — 50 Units
  Arms: AbobotulinumtoxinA Placebo
Drug: Placebo — 20 Units
  Arms: OnabotulinumtoxinA Placebo

SUMMARY:
The objective of this study is to demonstrate the efficacy of Dysport for the improvement in appearance of moderate to severe glabellar lines and to assess the short term and long term safety of Dysport, used for the improvement in appearance of moderate to severe glabellar lines in Chinese subjects.

DETAILED DESCRIPTION:
The first treatment cycle will be double blind and subjects will be randomised to receive Dysport, Botox or placebo. After the first treatment cycle, all subjects will receive a maximum of four treatment cycles with Dysport, occurring at intervals of no less than 84 Days (12 weeks) between each treatment cycle, depending upon individual duration of response to Dysport treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Male or female Chinese subjects who are between 18 to 65 years of age inclusive.
* Have moderate or severe wrinkles of vertical glabellar lines (Grade 2 or 3) at maximum frown at baseline (Day 1), as assessed by the subject using SSA.
* Have moderate or severe (Grade 2 or 3) vertical glabellar lines at maximum frown at baseline (Day 1), as assessed by the Investigator using ILA.
* Be Botulinum Toxin (BTX) naïve or have received their most recent BTX-A treatment more than 1 year prior to screening.
* Have a negative pregnancy test
* Have an understanding of the study

Exclusion Criteria:

* Any prior surgery affecting corrugator supercilii, prior blepharoplasty or brow lift, dermal resurfacing, or any prior cosmetic procedures or scars within 36 months.
* Any prior treatment with permanent fillers in the upper face.
* Any prior treatment with nonpermanent dermal fillers in the upper face within the past 3 years and/or skin abrasions/resurfacing, photorejuvenation or skin/vascular laser intervention within the past 12 months.
* Any planned facial cosmetic surgery or procedures during the study period.
* Lack of capacity to frown.
* Facial conditions that could affect safety or efficacy results.
* History of facial nerve palsy.
* Marked asymmetry; ptosis; excessive dermatochalasis; deep dermal scarring; thick sebaceous skin; photodamage etc.
* Presence of any condition that could affect the safety, conduct or outcome of the study.
* Any subjects who have any psychiatric illness or are taking antidepressant, anxiolytic or antipsychotic medication.
* Pregnant and/or lactating female subjects.
* Female subjects of childbearing potential not willing to use contraceptive measures throughout the course of the study.
* History of drug or alcohol abuse.
* Treatment with an experimental drug or device within 30 days prior to screening for this study and during the conduct of this study.
* Requirement for BTX injection to site(s) for disorders other than glabellar lines.
* Known allergy or hypersensitivity to BTX.
* Any medical condition or laboratory finding from central laboratory results.
* The subject is unable and/or unwilling to comply fully with the protocol and the study.
* Mental incapacity, unwillingness or language barriers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, M.D., Study Director — Ipsen
Locations (10):
- China (10):
  - Peking University First Hospital, Beijing
  - Air Force General Hospital, PLA, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The Third Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The Third Affiliated Hospital of Sun Yat-sen University, Guanzhou
  - Dermatology Hospital of the Chinese Academy of Medical Sciences, Nanjing
  - Tianjin Medical University General Hospital, Tianjing
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicentre, phase III, randomised, double-blind (DB) then open-label (OL) study. The 12 month recruitment period began in April 2015. A total of 555 subjects were screened across the 10 study centres in China and 520 subjects were randomised into the study.
Pre-assignment Details: The 35 screen failures were due to 17 subjects not meeting the eligibility criteria, 17 subjects withdrawing consent, and one subject reporting an adverse event.
Groups:
- Dysport® 50 Units (U) - DB Period: Subjects randomised to the Dysport® treatment group in Cycle 1 received on Day 1, 50 U (0.25 millilitres [mL]), divided into five injections into the glabellar area. 10 U (0.05 mL) of Dysport® was administered intramuscularly, at right angles to the skin into each of the five injection sites. The Investigator was blinded with respect to treatment injection.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57 and 85 of Cycle 1. On Day 85, subjects were assessed for their eligibility to enter the OL period (Cycles 2 to 5). Any subjects not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study. A subject was considered to have completed the study in Cycle 1 if they were not eligible for retreatment and had completed a total of 15 months follow-up following study treatment administration on Day 1.
- Dysport® Placebo - DB Period: Subjects randomised to the Dysport® placebo group in Cycle 1 received on Day 1, 0.25 mL, divided into five injections into the glabellar area. 0.05 mL of Dysport® placebo was administered intramuscularly, at right angles to the skin into each of the five injection sites. The Investigator was blinded with respect to treatment injection.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57 and 85 of Cycle 1. On Day 85, subjects were assessed for their eligibility to enter the OL period (Cycles 2 to 5). Any subjects not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study. A subject was considered to have completed the study in Cycle 1 if they were not eligible for retreatment and had completed a total of 15 months follow-up following study treatment administration on Day 1.
- Botox 20 U - DB Period: Subjects randomised to the Botox treatment group in Cycle 1 received on Day 1, 20 U (0.5 mL), divided into five injections into the glabellar area. 4 U (0.1 mL) of Botox was administered intramuscularly, at right angles to the skin into each of the five injection sites. The Investigator was blinded with respect to treatment injection.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57 and 85 of Cycle 1. On Day 85, subjects were assessed for their eligibility to enter the OL period (Cycles 2 to 5). Any subjects not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study. A subject was considered to have completed the study in Cycle 1 if they were not eligible for retreatment and had completed a total of 15 months follow-up following study treatment administration on Day 1.
- Botox Placebo - DB Period: Subjects randomised to the Botox placebo group in Cycle 1 received on Day 1, 0. 5 mL, divided into five injections into the glabellar area. 0.1 mL of Botox placebo was administered intramuscularly, at right angles to the skin into each of the five injection sites. The Investigator was blinded with respect to treatment injection.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57 and 85 of Cycle 1. On Day 85, subjects were assessed for their eligibility to enter the OL period (Cycles 2 to 5). Any subjects not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study. A subject was considered to have completed the study in Cycle 1 if they were not eligible for retreatment and had completed a total of 15 months follow-up following study treatment administration on Day 1.
- Dysport® 50 U - OL Period (Cycles 2-5): After the first treatment cycle, all eligible subjects entered the OL period and received Dysport® 50 U (0.25 mL), injected into five predefined sites across the glabellar region. 10 U (0.05 mL) of Dysport® was administered intramuscularly, at right angles to the skin into each of the five injection sites per treatment cycle.
  Subjects received a maximum of four treatment cycles (Cycles 2 to 5) with Dysport®. These cycles occurred at intervals of no less than 84 days (12 weeks) between each cycle, depending upon individual duration of response to Dysport® treatment. Any subjects not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study.
Period: DB Period (Cycle 1)
Arm/Group | Dysport® 50 Units (U) - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period | Dysport® 50 U - OL Period (Cycles 2-5)
Started (Subjects randomised to each treatment group.) | 325 | 66 | 107 | 22 | 0 (This arm was not included in DB Period (Cycle 1).)
Safety Population (1 subject was randomised to Botox placebo group but received treatment of Dysport® 50 U in Cycle 1.) | 326 | 66 | 107 | 21 | 0
Completed | 294 | 63 | 97 | 20 | 0 (This arm was not included in DB Period (Cycle 1).)
Not Completed | 31 | 3 | 10 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 28 | 3 | 8 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 1 | 0
Period: OL Period (Cycles 2-5)
Arm/Group | Dysport® 50 Units (U) - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period | Dysport® 50 U - OL Period (Cycles 2-5)
Started | 0 (This arm was not included in OL Period (Cycles 2-5).) | 0 (This arm was not included in OL Period (Cycles 2-5).) | 0 (This arm was not included in OL Period (Cycles 2-5).) | 0 (This arm was not included in OL Period (Cycles 2-5).) | 465 (Nine subjects completed the DB Period but were not eligible for retreatment in the OL Period.)
Safety Population | 0 | 0 | 0 | 0 | 465
Discontinued During Cycle 2 | 0 | 0 | 0 | 0 | 28
Discontinued During Cycle 3 | 0 | 0 | 0 | 0 | 11
Discontinued During Cycle 4 | 0 | 0 | 0 | 0 | 2
Discontinued During Cycle 5 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 424
Not Completed | 0 | 0 | 0 | 0 | 41
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 31
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Dysport® 50 U - DB Period: Subjects randomised to the Dysport® treatment group in Cycle 1 received on Day 1, 50 U (0.25 mL), divided into five injections into the glabellar area. 10 U (0.05 mL) of Dysport® was administered intramuscularly, at right angles to the skin into each of the five injection sites. The Investigator was blinded with respect to treatment injection.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57 and 85 of Cycle 1. On Day 85, subjects were assessed for their eligibility to enter the OL period (Cycles 2 to 5). Any subjects not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study. A subject was considered to have completed the study in Cycle 1 if they were not eligible for retreatment and had completed a total of 15 months follow-up following study treatment administration on Day 1.
- Total: Total of all reporting groups
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period | Total
Number analyzed (Participants) | 325 | 66 | 107 | 22 | 520
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 325 | 66 | 107 | 22 | 520
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (9.4) | 44.3 (9.5) | 44.9 (8.2) | 42.8 (9.8) | 45.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 57 | 94 | 19 | 452
  Male | 43 | 9 | 13 | 3 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 325 | 66 | 107 | 22 | 520
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Superiority Analysis of The Percentage of Responders Measured by the Investigator's Live Assessment (ILA) at Maximum Frown at Cycle 1, Day 29 (DB Period).
Description: At baseline (Cycle 1, Day 1) and at Cycle 1, Day 29, the Investigator assessed the appearance of the glabellar lines at maximum frown using a validated 4-point Photographic Scale of Glabellar Line Severity. This 4-point scale rated the severity of glabellar lines as Grade 0 (none), Grade 1 (mild), Grade 2 (moderate) and Grade 3 (severe). A responder was defined as having a severity grade of 0 or 1 at Cycle 1, Day 29, and a severity grade of 2 or 3 at maximum frown at baseline.
  Superiority analysis of active treatment versus placebo was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for Cycle 1, Day 29.
Time Frame: At Cycle 1, Day 29.
Population: The modified Intent-to-treat (mITT) population was all randomised subjects who received study treatment in at least one injection site regardless of the amount administered and had both the baseline and Cycle 1, Day 29 assessments, for the ILA and subjects' self assessment (SSA) of glabellar lines at maximum frown.
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
adjusted percentage of responders | 95.2 [91.2 to 97.4] | 0.9 [0.1 to 7.0] | 94.0 [85.2 to 97.7] | 4.3 [0.5 to 26.8]
Statistical Analysis 1: Comparison: Dysport® 50 U - DB Period vs Dysport® Placebo - DB Period; Superiority analysis of Dysport® to placebo was tested using a multivariate logistic regression model; Test type: Superiority — The model includes treatment group, stratification factors, gender and baseline severity score of glabellar lines at maximum frown measured by the ILA, and centre as explanatory variables and responder (Yes or No) as response variable; p < 0.0001, Regression, Logistic — The test is two-sided at the significance level of 0.025; Treatment difference = 94.3, 95% CI 2-sided [90.8 to 97.7]

2. Primary Outcome: Superiority Analysis of The Percentage of Responders Measured by the SSA at Maximum Frown at Cycle 1, Day 29 (DB Period).
Description: At baseline (Cycle 1, Day 1) and at Cycle 1, Day 29, subjects assessed the appearance of their glabellar lines at maximum frown using a 4-point categorical scale. The 4-point scale represents the severity of glabellar lines as Grade 0 (no wrinkles), Grade 1 (mild wrinkles), Grade 2 (moderate wrinkles) and Grade 3 (severe wrinkles). For the SSA, a responder was defined as having a severity grade of 0 or 1 at maximum frown at Cycle 1, Day 29, and a severity grade of 2 or 3 at maximum frown at baseline.
  Superiority analysis of active treatment versus placebo was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for Cycle 1, Day 29.
Time Frame: At Cycle 1, Day 29.
Population: The mITT population was all randomised subjects who received study treatment in at least one injection site regardless of the amount administered and had both the baseline and Cycle 1, Day 29 assessments, for the ILA and SSA of glabellar lines at maximum frown.
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
adjusted percentage of responders | 89.4 [84.4 to 93.0] | 1.9 [0.4 to 8.4] | 89.3 [79.2 to 94.9] | 1.5 [0.1 to 21.0]
Statistical Analysis 1: Comparison: Dysport® 50 U - DB Period vs Dysport® Placebo - DB Period; Superiority analysis of Dysport® to placebo was tested using a multivariate logistic regression model; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic — The test is two-sided at the significance level of 0.025; Treatment difference = 87.5, 95% CI 2-sided [82.5 to 92.4]

3. Primary Outcome: Non-Inferiority Analysis of The Percentage of Responders Measured by the Investigator's Live Assessment (ILA) at Maximum Frown at Cycle 1, Day 29 (DB Period).
Description: At baseline (Cycle 1, Day 1) and at Cycle 1, Day 29, the Investigator assessed the appearance of the glabellar lines at maximum frown using a validated 4-point Photographic Scale of Glabellar Line Severity. This 4-point scale rated the severity of glabellar lines as Grade 0 (none), Grade 1 (mild), Grade 2 (moderate) and Grade 3 (severe). A responder was defined as having a severity grade of 0 or 1 at Cycle 1, Day 29, and a severity grade of 2 or 3 at maximum frown at baseline.
  Non Inferiority analysis of Dysport® versus Botox was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for Cycle 1, Day 29.
Time Frame: At Cycle 1, Day 29.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Botox 20 U - DB Period
Number analyzed (Participants) | 294 | 94
adjusted percentage of responders | 94.7 [90.8 to 96.9] | 97.0 [92.0 to 98.9]
Statistical Analysis 1: Comparison: Dysport® 50 U - DB Period vs Botox 20 U - DB Period; The non-inferiority of Dysport® to Botox on the ILA at maximum frown was tested using a multivariate logistic regression model; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Treatment Difference = -2.4, 95% CI 2-sided [-6.7 to 1.9]

4. Secondary Outcome: The Percentage of Responders With Respect to Independent Reviewer's Assessment of Photographs of the Subject's Glabellar Lines at Maximum Frown at Cycle 1, Day 29 (DB Period).
Description: Photographs of the glabellar region of subjects were taken at maximum frown at baseline (Cycle 1, Day 1) and at Cycle 1, Day 29. Photographs were assessed by an Independent Experts Committee using a validated 4-point Photographic Scale of Glabellar Line Severity which rated the severity of glabellar lines as Grade 0 (none), Grade 1 (mild), Grade 2 (moderate) and Grade 3 (severe). The median of three readings by three independent reviewers was used in the analysis. A responder was defined as having a severity grade of 0 or 1 at Cycle 1, Day 29, and a severity grade of 2 or 3 at baseline.
  Superiority analysis of active treatment to placebo was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for Cycle 1, Day 29.
Time Frame: At Cycle 1, Day 29.
Population: The mITT population was all randomised subjects who received study treatment in at least one injection site regardless of the amount administered and had both the baseline and Cycle 1, Day 29 assessments, for the ILA and SSA of glabellar lines at maximum frown. Subjects with a baseline score of 0 or 1 are excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 194 | 34 | 60 | 11
adjusted percentage of responders | 99.1 [95.0 to 99.8] | 25.3 [11.6 to 46.7] | 94.4 [85.0 to 98.1] | 31.5 [9.4 to 67.1]
Statistical Analysis 1: Comparison: Dysport® 50 U - DB Period vs Dysport® Placebo - DB Period; Superiority analysis of Dysport® to placebo was tested using a multivariate logistic regression model; Test type: Superiority — The model includes treatment group, stratification factors, gender and baseline severity score of glabellar lines at maximum frown measured by the ILA and centre as explanatory variables and responder (Yes or No) as response variable; p < 0.0001, Regression, Logistic; Treatment difference = 73.8, 95% CI 2-sided [59.1 to 88.4]

5. Secondary Outcome: Mean Subject's Global Assessment (SGA) Score at Cycle 1, Day 29 (DB Period).
Description: On Cycle 1, Day 29, subjects were asked to assess the change, since the last treatment administration, in the appearance of their glabellar lines using the following 9-point Global Assessment Scale: +4 =100% improvement; +3 =75% improvement; +2 =50% improvement; +1 =25% improvement; 0 =no change; -1 =25% worsening; -2 =50%worsening; -3 =75% worsening; -4 =100% worsening.
  The mean SGA score at Cycle 1, Day 29 is presented.
Time Frame: At Cycle 1, Day 29.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on the SGA scale
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
units on the SGA scale | 2.6 (1.1) | 0.1 (0.4) | 2.7 (1.1) | 0.1 (0.3)
Statistical Analysis 1: Comparison: Dysport® 50 U - DB Period vs Dysport® Placebo - DB Period; Superiority analysis of Dysport® to placebo was tested using a linear mixed model; Test type: Superiority — The comparison between mean scores of SGA at Treatment Cycle 1, Day 29 is based on 2 separate linear mixed models, adjusting on the two stratification parameters, gender and baseline ILA severity score, and the centre; p < 0.0001, Mixed Models Analysis — The test was two-sided at the significance level of 0.05; Treatment Difference = 2.603, 95% CI 2-sided [2.327 to 2.878]

6. Secondary Outcome: The Percentage of Responders With Respect to the SGA Score at Cycle 1, Day 29 (DB Period).
Description: On Cycle 1, Day 29, subjects were asked to assess the change, since the last treatment administration, in the appearance of their glabellar lines using the following 9-point Global Assessment Scale: +4 =100% improvement; +3 =75% improvement; +2 =50% improvement; +1 =25% improvement; 0 =no change; -1 =25% worsening; -2 =50% worsening; -3 =75% worsening; -4 =100% worsening. A responder, based on the SGA scale, was defined as having a grade of at least +2 (50% improvement).
  Superiority analysis of active treatment versus placebo was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for Cycle 1, Day 29.
Time Frame: At Cycle 1, Day 29.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
adjusted percentage of responders | 85.1 [80.2 to 88.9] | 1.3 [0.2 to 9.0] | 85.2 [74.4 to 91.9] | 2.4 [0.2 to 23.3]
Statistical Analysis 1: Comparison: Dysport® 50 U - DB Period vs Dysport® Placebo - DB Period; Superiority analysis of Dysport® to placebo was tested using a multivariate logistic regression model; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic; Treatment difference = 83.7, 95% CI 2-sided [78.7 to 88.7]

7. Other Pre Specified Outcome: The Percentage of Responders Measured by the ILA at Maximum Frown at Cycle 1 Study Visits (DB Period).
Description: At baseline (Cycle 1, Day 1) and at all subsequent study visits, the Investigator assessed the appearance of the glabellar lines at maximum frown using a validated 4-point photographic scale of glabellar line severity. This 4-point scale rated the severity of glabellar lines as Grade 0 (none), Grade 1 (mild), Grade 2 (moderate) and Grade 3 (severe). A responder was defined as having a severity grade of 0 or 1 at any given visit, and a severity grade of 2 or 3 at baseline.
  Superiority analysis of active treatment versus placebo was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for all visits up to Day 85 in the DB period (except Cycle 1, Day 29).
Time Frame: Up to Cycle 1, Day 85.
Population: The mITT population was all randomised subjects who received study treatment in at least one injection site regardless of the amount administered and had both the baseline and Cycle 1, Day 29 assessments, for the ILA and SSA of glabellar lines at maximum frown. Only subjects with data available for analysis at each time point are presented.
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
adjusted percentage of responders
  Cycle 1, Day 8 | 86.3 [81.0 to 90.3] | 1.0 [0.1 to 6.9] | 87.3 [76.1 to 93.7] | 1.1 [0.1 to 18.4]
  Cycle 1, Day 57 | 87.7 [82.7 to 91.4] | 2.9 [0.8 to 9.7] | 92.6 [79.4 to 97.6] | 1.0 [0.0 to 20.7]
  Cycle 1, Day 85 | 80.3 [72.1 to 86.6] | 0.1 [0.0 to 3.2] | 76.4 [63.8 to 85.6] | 1.1 [0.0 to 22.4]

8. Other Pre Specified Outcome: The Percentage of Responders Measured by the SSA at Maximum Frown at Cycle 1 Study Visits (DB Period).
Description: At baseline (Cycle 1, Day 1) and all subsequent study visits, subjects assessed the appearance of their glabellar lines at maximum frown using a 4-point categorical scale. The 4-point scale represents the severity of glabellar lines as Grade 0 (no wrinkles), Grade 1 (mild wrinkles), Grade 2 (moderate wrinkles) and Grade 3 (severe wrinkles). For the SSA, a responder was defined as having a severity grade of 0 or 1 at maximum frown at any given visit, and a severity grade of 2 or 3 at maximum frown at baseline.
  Superiority analysis of active treatment versus placebo was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for all visits up to Day 85 in the DB period (except Cycle 1, Day 29).
Time Frame: Up to Cycle 1, Day 85.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
adjusted percentage of responders
  Cycle 1, Day 8 | 78.6 [72.7 to 83.5] | 2.0 [0.5 to 8.5] | 77.3 [66.4 to 85.5] | 7.4 [1.5 to 29.8]
  Cycle 1, Day 57 | 84.9 [79.6 to 89.0] | 2.1 [0.5 to 8.7] | 88.1 [76.8 to 94.4] | 2.6 [0.2 to 23.5]
  Cycle 1, Day 85 | 68.2 [61.5 to 74.2] | 1.7 [0.4 to 7.1] | 72.2 [59.4 to 82.3] | 1.0 [0.0 to 21.5]

9. Other Pre Specified Outcome: The Percentage of Responders Measured by the ILA at Rest at Cycle 1 Study Visits (DB Period).
Description: At baseline (Cycle 1, Day 1) and at all subsequent study visits, the Investigator assessed the appearance of the glabellar lines at rest using a validated 4-point photographic scale of glabellar line severity. This 4-point scale rated the severity of glabellar lines as Grade 0 (none), Grade 1 (mild), Grade 2 (moderate) and Grade 3 (severe). A responder was defined as having a severity grade of 0 or 1 at rest at any given visit, and a severity grade of 2 or 3 at rest at baseline.
  Superiority analysis of active treatment versus placebo was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for all visits up to Day 85 in the DB period (except Cycle 1, Day 29).
Time Frame: Up to Cycle 1, Day 85.
Population: The mITT population was all randomised subjects who received study treatment in at least one injection site regardless of the amount administered and had both the baseline and Cycle 1, Day 29 assessments, for the ILA and SSA of glabellar lines at maximum frown. Subjects with a baseline score of 0 or 1 were excluded from the analysis of responders.
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 123 | 17 | 33 | 3
adjusted percentage of responders
  Cycle 1, Day 8 | 54.2 [44.4 to 63.6] | 12.2 [2.8 to 39.6] | 65.4 [44.4 to 81.7] | 8.4 [0.2 to 82.2]
  Cycle 1, Day 57 | 66.5 [55.6 to 75.9] | 13.1 [3.2 to 40.5] | 68.2 [47.3 to 83.7] | 24.9 [1.5 to 87.7]
  Cycle 1, Day 85 | 61.8 [51.1 to 71.4] | 22.1 [7.4 to 50.1] | 71.8 [49.3 to 87.0] | 5.8 [0.1 to 75.0]

10. Other Pre Specified Outcome: The Percentage of Responders With Respect to Independent Reviewer's Assessment of Photographs of the Subject's Glabellar Lines at Maximum Frown at Cycle 1, Day 85 (DB Period).
Description: Photographs of the glabellar region of subjects were taken at baseline and at maximum frown at Cycle 1, Day 85. Photographs were assessed by an Independent Experts Committee using a validated 4-point Photographic Scale of Glabellar Line Severity. This 4-point scale rated the severity of glabellar lines as Grade 0 (none), Grade 1 (mild), Grade 2 (moderate) and Grade 3 (severe). The median of 3 readings by 3 independent reviewers was used in the analysis. A responder was defined as having a severity grade of 0 or 1 at Cycle 1, Day 85, and a severity grade of 2 or 3 at baseline.
  Superiority analysis of active treatment versus placebo was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for Cycle 1, Day 85 .
Time Frame: At Cycle 1, Day 85.
Population: The mITT population was all randomised subjects who received study treatment in at least one injection site regardless of the amount administered and had both the baseline and Cycle 1, Day 29 assessments, for the ILA and SSA of glabellar lines at maximum frown. Subjects with a baseline score of 0 or 1 were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
adjusted percentage of responders | 93.3 [87.4 to 96.5] | 13.5 [5.1 to 30.9] | 89.0 [74.5 to 95.7] | 22.0 [5.6 to 57.0]

11. Other Pre Specified Outcome: Mean SGA Score at Cycle 1 Study Visits (DB Period).
Description: On all study visits, subjects were asked to assess the change, since the last treatment administration, in the appearance of their glabellar lines using the following 9-point Global Assessment Scale: +4 =100% improvement; +3 =75% improvement; +2 =50% improvement; +1 =25% improvement; 0 =no change; -1 =25% worsening; -2 =50% worsening; -3 =75% worsening; -4 =100% worsening.
  The mean SGA score for study visits on Day 8 to Day 85 in the DB period is presented (except Cycle 1, Day 29).
Time Frame: Up to Cycle 1, Day 85.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on the SGA scale
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
units on the SGA scale
  Cycle 1, Day 8 | 2.3 (1.2) | 0.1 (0.4) | 2.3 (1.3) | 0.2 (0.5)
  Cycle 1, Day 57: number analyzed (Participants) | 293 | 59 | 94 | 18
  Cycle 1, Day 57 | 2.4 (1.2) | 0.1 (0.6) | 2.4 (1.1) | 0.1 (0.4)
  Cycle 1, Day 85: number analyzed (Participants) | 294 | 59 | 94 | 18
  Cycle 1, Day 85 | 1.9 (1.3) | 0.1 (0.6) | 1.8 (1.2) | 0.1 (0.2)

12. Other Pre Specified Outcome: The Percentage of Responders With Respect to the SGA Score at Cycle 1 Study Visits (DB Period).
Description: On all study visits, subjects were asked to assess the change, since the last treatment administration, in the appearance of their glabellar lines using the following 9-point Global Assessment Scale: +4 =100% improvement; +3 =75% improvement; +2 =50% improvement; +1 =25% improvement; 0 =no change; -1 =25% worsening; -2 =50%worsening; -3 =75% worsening; -4 =100% worsening. A responder, based on the SGA scale, was defined as having a grade of at least +2 (50% improvement).
  Superiority analysis of active treatment versus placebo was carried out using a multivariate logistic regression model and adjusted for the stratification factors of gender and baseline severity score of glabellar lines at maximum frown measured by the ILA. The adjusted percentage of responders is presented for all visits up to Day 85 in the DB period (except Cycle 1, Day 29).
Time Frame: Up to Cycle 1, Day 85.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: adjusted percentage of responders
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
adjusted percentage of responders
  Cycle 1, Day 8 | 78.0 [72.3 to 82.7] | 1.2 [0.2 to 8.5] | 73.7 [62.5 to 82.5] | 2.8 [0.3 to 22.8]
  Cycle 1, Day 57 | 80.1 [74.4 to 84.7] | 3.4 [1.0 to 10.7] | 79.5 [67.8 to 87.8] | 1.8 [0.1 to 22.2]
  Cycle 1, Day 85 | 65.2 [59.1 to 70.9] | 2.5 [0.6 to 9.7] | 57.4 [46.5 to 67.5] | 2.0 [0.1 to 23.5]

13. Other Pre Specified Outcome: Least Squares (LS) Mean Change From Baseline in Subject's Self-perception of Age at Cycle 1 Study Visits (DB Period).
Description: At baseline (Cycle 1, Day 1) and all subsequent study visits in Cycle 1, subjects were asked to evaluate their age over the past 7 days at the time of assessment, using the following categories:
  * I look like my current age;
  * I look _ years younger;
  * I look _ years older.
  The LS mean change from baseline in subject's self-perception of age at all study visits in the DB Period was calculated. A negative LS mean change from baseline in the subject's self-perception of age indicates that the subject's self-perception was to look younger compared with baseline.
Time Frame: Up to Cycle 1, Day 85.
Population: The mITT population was all randomised subjects who received study treatment in at least one injection site regardless of the amount administered and had both the baseline and Cycle 1, Day 29 assessments, for the ILA and SSA of glabellar lines at maximum frown. Only subjects with data available for analysis at each time point is presented.
Measure: Least Squares Mean (Standard Error); unit: years
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 294 | 60 | 94 | 19
years
  Cycle 1, Day 8 | -2.083 (0.278) | 0.344 (0.471) | -1.442 (0.422) | -0.266 (0.710)
  Cycle 1, Day 29 | -2.566 (0.296) | 0.478 (0.524) | -2.421 (0.437) | -0.003 (0.754)
  Cycle 1, Day 57: number analyzed (Participants) | 293 | 59 | 94 | 18
  Cycle 1, Day 57 | -2.483 (0.293) | 0.698 (0.515) | -1.857 (0.420) | -0.453 (0.711)
  Cycle 1, Day 85: number analyzed (Participants) | 290 | 58 | 93 | 18
  Cycle 1, Day 85 | -2.035 (0.281) | 0.581 (0.481) | -1.374 (0.452) | -0.208 (0.802)

14. Other Pre Specified Outcome: The Time to Onset of Treatment Response Based on the Subject's Diary Card (DB Period).
Description: Subjects were given the diary card at baseline (Cycle 1, Day 1 ) and asked to record their assessment of study treatment response for the first 7 days post-treatment (Days 2 to 8). They were asked to respond 'yes' or 'no' to the following question: 'Since being injected have you noticed an improvement in the appearance of your glabellar lines (lines between your eyebrows)?' Subjects with no treatment response were censored at the date of last assessment of treatment response recorded in the diary card.
  The 50th percentile of Kaplan-Meier estimates was used to estimate the median time to onset of treatment response for each treatment group.
Time Frame: At Cycle 1, Day 8.
Population: The mITT population was all randomised subjects who received study treatment in at least one injection site regardless of the amount administered and had both the baseline and Cycle 1, Day 29 assessments, for the ILA and SSA of glabellar lines at maximum frown. Only subjects with treatment response on Cycle 1, Day 8 were analysed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period
Number analyzed (Participants) | 268 | 8 | 82 | 5
days | 2.0 [2.0 to 3.0] | NA [NA to NA] — Results were non-calculable due to censored data. | 3.0 [2.0 to 3.0] | NA [7.0 to NA] — Results were non-calculable due to censored data.

15. Other Pre Specified Outcome: The Percentage of Responders Measured by the ILA at Maximum Frown at All Other Study Visits (OL Period).
Description: At baseline (Cycle 1, Day 1) and all subsequent study visits (per treatment cycle) in the OL period, the Investigator assessed the appearance of the glabellar lines at maximum frown using a validated 4-point Photographic Scale of Glabellar Line Severity. This 4-point scale rated the severity of glabellar lines as Grade 0 (none), Grade 1 (mild), Grade 2 (moderate) and Grade 3 (severe). A responder was defined as having a severity grade of 0 or 1 at each study visit, and a severity grade of 2 or 3 at baseline.
  The proportion (percentage) of responders measured by ILA at all study visits in each treatment cycle, is presented.
Time Frame: Up to Cycle 5, Day 85.
Population: The OL population was all randomised subjects who received any dose of OL Dysport®. Only subjects with data available for analysis at each time point are presented.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- Dysport® 50 U, Cycle 2 (OL Period): All subjects who were eligible for retreatment following the DB period entered Cycle 2 and received OL Dysport® 50 U. The total treatment dose was injected in 5 predefined sites across the glabellar region on Cycle 2, Day 1.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57, and 85 of Cycle 2. Subjects were assessed for the eligibility to receive the next treatment cycle from Day 85.
  Any subjects who were not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study. A subject was considered to have completed the study when they had either received a total of five study treatment injections or completed a total of 15 months follow-up in the study following the first study treatment administration and completed the Day 85 visit following the last injection.
- Dysport® 50 U, Cycle 3 (OL Period): All subjects who were eligible for retreatment following Cycle 2 entered Cycle 3 and received OL Dysport® 50 U. The total treatment dose was injected in 5 predefined sites across the glabellar region on Cycle 3 Day 1.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57, and 85 of Cycle 3. Subjects were assessed for the eligibility to receive the next treatment cycle from Day 85.
  Any subjects who were not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study. A subject was considered to have completed the study when they had either received a total of five study treatment injections or completed a total of 15 months follow-up in the study following the first study treatment administration and completed the Day 85 visit following the last injection.
- Dysport® 50 U, Cycle 4 (OL Period): All subjects who were eligible for retreatment following Cycle 3 entered Cycle 4 and received OL Dysport® 50 U. The total treatment dose was injected in 5 predefined sites across the glabellar region on Cycle 4, Day 1.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57, and 85 of Cycle 4. Subjects were assessed for the eligibility to receive the next treatment cycle from Day 85.
  Any subjects who were not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study. A subject was considered to have completed the study when they had either received a total of five study treatment injections or completed a total of 15 months follow-up in the study following the first study treatment administration and completed the Day 85 visit following the last injection.
- Dysport® 50 U, Cycle 5 (OL Period): All subjects who were eligible for retreatment following Cycle 4 entered Cycle 5 and received OL Dysport® 50 U. The total treatment dose was injected in 5 predefined sites across the glabellar region on Cycle 5, Day 1.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57, and 85 of Cycle 5. A subject was considered to have completed the study when they had either received a total of five study treatment injections or completed a total of 15 months follow-up in the study following the first study treatment administration and completed the Day 85 visit following the last injection.
Arm/Group | Dysport® 50 U, Cycle 2 (OL Period) | Dysport® 50 U, Cycle 3 (OL Period) | Dysport® 50 U, Cycle 4 (OL Period) | Dysport® 50 U, Cycle 5 (OL Period)
Number analyzed (Participants) | 424 | 355 | 232 | 98
percentage of responders
  Day 8: number analyzed (Participants) | 422 | 350 | 227 | 96
  Day 8 | 92.9 [90.1 to 95.2] | 92.1 [88.8 to 94.7] | 92.2 [88.0 to 95.3] | 84.7 [76.0 to 91.2]
  Day 29: number analyzed (Participants) | 410 | 348 | 226 | 97
  Day 29 | 92.7 [89.8 to 95.0] | 93.5 [90.4 to 95.8] | 90.1 [85.5 to 93.6] | 84.7 [76.0 to 91.2]
  Day 57: number analyzed (Participants) | 410 | 349 | 227 | 97
  Day 57 | 88.0 [84.5 to 90.9] | 88.7 [85.0 to 91.8] | 85.8 [80.6 to 90.0] | 81.6 [72.5 to 88.7]
  Day 85: number analyzed (Participants) | 407 | 348 | 231 | 98
  Day 85 | 71.7 [67.2 to 75.9] | 73.8 [68.9 to 78.3] | 68.1 [61.7 to 74.1] | 61.2 [50.8 to 70.9]

16. Other Pre Specified Outcome: The Percentage of Responders Measured by the SSA at Maximum Frown at All Other Study Visits (OL Period).
Description: At baseline (Cycle 1, Day 1) and all subsequent study visits per treatment cycle in the OL period, subjects assessed the appearance of their glabellar lines at maximum frown using a 4-point categorical scale. The 4-point scale represents the severity of glabellar lines as Grade 0 (no wrinkles), Grade 1 (mild wrinkles), Grade 2 (moderate wrinkles) and Grade 3 (severe wrinkles). For the SSA, a responder was defined as having a severity grade of no wrinkles (0) or mild wrinkles (1) at maximum frown at a given visit and a severity grade of moderate wrinkles (2) or severe wrinkles (3) at maximum frown at baseline.
  The proportion (percentage) of responders measured by SSA at all study visits in Cycle 2 to 5 is presented.
Time Frame: Up to Cycle 5, Day 85.
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Dysport® 50 U, Cycle 2 (OL Period) | Dysport® 50 U, Cycle 3 (OL Period) | Dysport® 50 U, Cycle 4 (OL Period) | Dysport® 50 U, Cycle 5 (OL Period)
Number analyzed (Participants) | 424 | 355 | 232 | 98
percentage of responders
  Day 8: number analyzed (Participants) | 422 | 349 | 227 | 96
  Day 8 | 85.3 [81.6 to 88.6] | 89.0 [85.3 to 92.1] | 87.5 [82.5 to 91.5] | 77.6 [68.0 to 85.4]
  Day 29: number analyzed (Participants) | 411 | 348 | 226 | 97
  Day 29 | 89.1 [85.8 to 91.9] | 88.5 [84.7 to 91.6] | 87.5 [82.5 to 91.5] | 77.6 [68.0 to 85.4]
  Day 57: number analyzed (Participants) | 410 | 349 | 227 | 97
  Day 57 | 85.1 [81.4 to 88.4] | 83.9 [79.7 to 87.6] | 82.8 [77.3 to 87.4] | 71.4 [61.4 to 80.1]
  Day 85: number analyzed (Participants) | 406 | 348 | 231 | 98
  Day 85 | 68.8 [64.1 to 73.2] | 70.7 [65.7 to 75.4] | 62.5 [55.9 to 68.7] | 62.2 [51.9 to 71.8]

17. Other Pre Specified Outcome: The Percentage of Responders Measured by the ILA at Rest at All Study Visits (OL Period).
Description: At baseline (Cycle 1, Day 1) and all subsequent study visits per treatment cycle in the OL period, the Investigator assessed the appearance of the glabellar lines at rest using a validated 4-point Photographic Scale of Glabellar Line Severity. This 4-point scale rated the severity of glabellar lines as Grade 0 (none), Grade 1 (mild), Grade 2 (moderate) and Grade 3 (severe). A responder was defined as having a severity grade of 0 or 1 at a given visit, and a severity grade of 2 or 3 at baseline. Subjects with a baseline score of 0 or 1 were excluded from the analysis of responders. The proportion (percentage) of responders measured by ILA at all study visits per treatment cycle in in the OL period is presented.
Time Frame: Up to Cycle 5, Day 85.
Population: The OL population was all randomised subjects who received any dose of OL Dysport®. Only subjects with a baseline score of 2 or 3 and with data available for analysis at each time point are presented.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Dysport® 50 U, Cycle 2 (OL Period) | Dysport® 50 U, Cycle 3 (OL Period) | Dysport® 50 U, Cycle 4 (OL Period) | Dysport® 50 U, Cycle 5 (OL Period)
Number analyzed (Participants) | 109 | 69 | 44 | 16
percentage of responders
  Day 8 | 60.6 [50.7 to 69.8] | 52.2 [39.8 to 64.4] | 54.5 [38.8 to 69.6] | 18.8 [4.0 to 45.6]
  Day 29 | 63.3 [53.5 to 72.3] | 58.0 [45.5 to 69.8] | 54.5 [38.8 to 69.6] | 25.0 [7.3 to 52.4]
  Day 57 | 62.4 [52.6 to 71.5] | 56.5 [44.0 to 68.4] | 54.5 [38.8 to 69.6] | 25.0 [7.3 to 52.4]
  Day 85 | 56.9 [47.0 to 66.3] | 58.0 [45.5 to 69.8] | 59.1 [43.2 to 73.7] | 25.0 [7.3 to 52.4]

18. Other Pre Specified Outcome: Mean SGA Score at All Other Study Visits (OL Period).
Description: On each study visit per treatment cycle in the OL period, subjects were asked to assess the change, since the last treatment administration, in the appearance of their glabellar lines using the following 9-point Global Assessment Scale: +4 =100% improvement; +3 =75% improvement; +2 =50% improvement; +1 =25% improvement; 0 =no change; -1 =25% worsening; -2 =50%worsening; -3 =75% worsening; -4 =100% worsening.
  The mean SGA score for study visits on Day 8 to Day 85 in the OL period is presented.
Time Frame: Up to Cycle 5, Day 85.
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on the SGA scale
Arm/Group | Dysport® 50 U, Cycle 2 (OL Period) | Dysport® 50 U, Cycle 3 (OL Period) | Dysport® 50 U, Cycle 4 (OL Period) | Dysport® 50 U, Cycle 5 (OL Period)
Number analyzed (Participants) | 424 | 355 | 232 | 98
units on the SGA scale
  Day 8: number analyzed (Participants) | 422 | 350 | 227 | 98
  Day 8 | 2.5 (1.1) | 2.4 (1.1) | 2.5 (1.2) | 2.1 (1.1)
  Day 29: number analyzed (Participants) | 410 | 348 | 226 | 97
  Day 29 | 2.6 (1.1) | 2.5 (1.0) | 2.4 (1.1) | 2.1 (1.2)
  Day 57: number analyzed (Participants) | 410 | 349 | 227 | 97
  Day 57 | 2.4 (1.1) | 2.3 (1.2) | 2.2 (1.1) | 1.9 (1.1)
  Day 85: number analyzed (Participants) | 406 | 348 | 231 | 98
  Day 85 | 2.0 (1.2) | 1.9 (1.2) | 1.8 (1.2) | 1.5 (1.2)

19. Other Pre Specified Outcome: The Proportion of Responders With Respect to the SGA Score at All Other Study Visits (OL Period).
Description: On each study visit per treatment cycle in the OL period, subjects were asked to assess the change, since the last treatment administration, in the appearance of their glabellar lines using the following 9-point Global Assessment Scale: +4 =100% improvement; +3 =75% improvement; +2 =50% improvement; +1 =25% improvement; 0 =no change; -1 =25% worsening; -2 =50%worsening; -3 =75% worsening; -4 =100% worsening.
  A responder, based on the SGA scale, was defined as having a grade of at least +2 (50% improvement). The proportion (percentage) of responders at each study visit on Day 8 to Day 85 in the OL period is presented.
Time Frame: Up to Cycle 5, Day 85.
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Dysport® 50 U, Cycle 2 (OL Period) | Dysport® 50 U, Cycle 3 (OL Period) | Dysport® 50 U, Cycle 4 (OL Period) | Dysport® 50 U, Cycle 5 (OL Period)
Number analyzed (Participants) | 424 | 355 | 232 | 98
percentage of responders
  Day 8: number analyzed (Participants) | 422 | 350 | 227 | 96
  Day 8 | 81.4 [77.3 to 85.0] | 75.5 [70.7 to 79.9] | 76.3 [70.3 to 81.6] | 62.2 [51.9 to 71.8]
  Day 29: number analyzed (Participants) | 410 | 348 | 226 | 97
  Day 29 | 82.1 [78.1 to 85.6] | 80.3 [75.8 to 84.3] | 75.4 [69.4 to 80.8] | 65.3 [55.0 to 74.6]
  Day 57: number analyzed (Participants) | 410 | 349 | 227 | 97
  Day 57 | 77.4 [73.1 to 81.3] | 74.4 [69.5 to 78.8] | 70.3 [63.9 to 76.1] | 66.3 [56.1 to 75.6]
  Day 85: number analyzed (Participants) | 406 | 348 | 231 | 98
  Day 85 | 63.4 [58.7 to 68.0] | 65.4 [60.1 to 70.3] | 61.6 [55.0 to 67.9] | 52.0 [41.7 to 62.2]

20. Other Pre Specified Outcome: Mean Change From Baseline in Subject's Self-Perception of Age at All Study Visits (OL Period)
Description: At cycle baseline (Day 1 of each treatment cycle) and Day 29 of each cycle in the OL period, subjects were asked to evaluate their age over the past 7 days at the time of assessment, using the following categories:
  * I look like my current age;
  * I look _ years younger;
  * I look _ years older.
  The mean change from cycle baseline in subject's self-perception of age at Day 29 of each cycle of the OL Period was calculated. A negative mean change from baseline in the subject's self-perception of age indicates that the subject's self-perception was to look younger compared with baseline.
Time Frame: Up to Cycle 5, Day 29.
Population: The OL population was all randomised subjects who received any dose of OL Dysport®. Only subjects with data available for analysis is presented.
Measure: Mean (Standard Deviation); unit: years
Groups:
- Dysport® 50 U, Cycle 2 (OL Period): All subjects who were eligible for retreatment following the DB period entered Cycle 2 and received OL Dysport® 50 U. The total treatment dose was injected in 5 predefined sites across the glabellar region on Cycle 2 Day 1.
  Following treatment administration, all subjects attended follow-up visits on Days 8, 29, 57, and 85 of Cycle 2. Subjects were assessed for the eligibility to receive the next treatment cycle from Day 85.
  Any subjects who were not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study. A subject was considered to have completed the study when they had either received a total of five study treatment injections or completed a total of 15 months follow-up in the study following the first study treatment administration and completed the Day 85 visit following the last injection.
Arm/Group | Dysport® 50 U, Cycle 2 (OL Period) | Dysport® 50 U, Cycle 3 (OL Period) | Dysport® 50 U, Cycle 4 (OL Period) | Dysport® 50 U, Cycle 5 (OL Period)
Number analyzed (Participants) | 410 | 347 | 225 | 97
years | -1.9 (3.0) | -1.6 (2.9) | -1.6 (3.0) | -1.1 (2.4)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were defined as any adverse event with start date on or after the first injection of study treatment or with start date prior to the first injection of study treatment but the intensity increased after the first injection of study treatment. TEAEs were collected until the end of Cycle 5 of the OL period, over a total timeframe of up to approximately 29 months.
Description: The safety population consisted of all randomised subjects who received at least one injection of study treatment into at least one injection site. The safety population was analysed based on the treatment the subject actually received rather than the treatment to which the subject was randomised. The 1 subject who was randomised to Botox placebo group but received treatment of Dysport® 50 U in Cycle 1 was included in the Dysport® 50 U group and excluded from the Botox placebo group.
Groups:
- Dysport® 50 U - OL Period: After the first treatment cycle, all eligible subjects entered the OL period and received Dysport® 50 U (0.25 mL), injected into five predefined sites across the glabellar region. 10 U (0.05 mL) of Dysport® was administered intramuscularly, at right angles to the skin into each of the five injection sites per treatment cycle.
  Subjects received a maximum of four treatment cycles (Cycles 2 to 5) with Dysport®. These cycles occurred at intervals of no less than 84 days (12 weeks) between each cycle, depending upon individual duration of response to Dysport® treatment. Any subjects not eligible for retreatment were evaluated every 28 days at additional follow-up visits until they were eligible for retreatment or had completed the study
Arm/Group | Dysport® 50 U - DB Period | Dysport® Placebo - DB Period | Botox 20 U - DB Period | Botox Placebo - DB Period | Dysport® 50 U - OL Period
All-Cause Mortality (participants affected / at risk) | 0/326 | 0/66 | 0/107 | 0/21 | 0/465
Serious Adverse Events (participants affected / at risk) | 5/326 | 2/66 | 2/107 | 0/21 | 28/465
Other Adverse Events (participants affected / at risk) | 83/326 | 9/66 | 23/107 | 4/21 | 142/465
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® 50 U - DB Period (N=326) | Dysport® Placebo - DB Period (N=66) | Botox 20 U - DB Period (N=107) | Botox Placebo - DB Period (N=21) | Dysport® 50 U - OL Period (N=465)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrosalpinx (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® 50 U - DB Period (N=326) | Dysport® Placebo - DB Period (N=66) | Botox 20 U - DB Period (N=107) | Botox Placebo - DB Period (N=21) | Dysport® 50 U - OL Period (N=465)
Eyelid oedema (Eye disorders) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Eyelid ptosis (Eye disorders) | 13 (13) | 0 (0) | 1 (1) | 0 (0) | 15 (16)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 29 (35) | 4 (5) | 12 (13) | 0 (0) | 74 (94)
Viral upper respiratory tract infection (Infections and infestations) | 15 (18) | 3 (3) | 4 (4) | 0 (0) | 25 (27)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 9 (10) | 0 (0) | 1 (1) | 0 (0) | 9 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 6 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 10 (10)
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 12 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor must review all results communications prior to public release. The sponsor has the right to delay a publication by 60 days from the time submitted to the sponsor for review. Any factual amendments proposed by sponsor will be incorporated, provided that they do not alter the scientific value of the material.